CLINICAL TRIAL: NCT04041362
Title: A Phase II, Open-label, Controlled, Proof-of-concept Study to Evaluate the Safety of UB-421 in Combination With Antiretroviral Therapy (ART) and the Efficacy in Reduction of HIV Viral Load and Proviral DNA as Compared to ART Alone in ART-experienced Viremic HIV-1 Patients
Brief Title: the Study to Evaluate the Safety of UB-421 in Combination With Antiretroviral Therapy (ART) and the Efficacy in Reduction of HIV Viral Load and Proviral DNA as Compared to ART Alone in ART-experienced Viremic HIV-1 Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study will not be submitted to authority for IND application.
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A213-HIV
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2019-11

CONDITIONS: HIV-1 Infection
Keywords: HIV; UB-421
MeSH Terms: interventions — UB-421; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1 (Standard ART) (Active Comparator): Standard ART
  Interventions: Other: Antiretroviral Therapy (ART)
- Arm 2 (ART plus UB-421) (Experimental): ART plus weekly UB-421 IV infusion at 5 mg/kg dose level for 16 weeks
  Interventions: Biological: UB-421; Other: Antiretroviral Therapy (ART)

INTERVENTIONS:
Biological: UB-421 — Monoclonal antibody by IV infusion plus standard ART
  Arms: Arm 2 (ART plus UB-421)
Other: Antiretroviral Therapy (ART) — Standard ART

SUMMARY:
This study assess the safety, tolerability, and efficacy in reducing viral load and proviral DNA of UB-421 administered as an add-on to the ART in ART-experienced viremic HIV-1 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 seropositive
2. Male with body weight ≥ 50 kg or female with body weight ≥ 45 kg.
3. have been receiving antiretroviral therapy (ART) for more than 2 years

Exclusion Criteria:

1. Any previous exposure to a mAb within 12 weeks prior to the first dose of UB-421 treatment.
2. Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined during the screening period, medical history, and/or physical examination that, in Investigator's opinion, would preclude the subject from participating in this study.
3. History of anaphylaxis to monoclonal antibodies.
4. Any vaccination within 8 weeks prior to the first dose of UB-421.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
treatment related TEAEs | 16 Weeks
  the incidence of Grade 3 drug-related treatment-emergent adverse events

IPD SHARING:
Plan to Share IPD: No